CLINICAL TRIAL: NCT04710615
Title: Impact of an Artificial Intelligence Platform on Inappropriate Medication Use in Older Adults
Acronym: PING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2019/33
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Drug-drug Interactions; Geriatric Disease
Keywords: Drugs; artificial; intelligence; medications; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assistance device (Experimental): With prescription assistance device:
  During the other 3 months, investigators will have the Synapse platform on different media (mobile phones, tablets, laptops and landline).
  Interventions: Device: Synapse platform
- No device (No Intervention): During 3 months, investigators will not have the Synapse platform and will make their prescriptions with the usual tools which they have: Modules of help in the DxCare® software of the CHU, public database of the drugs, dictionary Vidal®, …

INTERVENTIONS:
Device: Synapse platform — The Synapse platform made available to health professionals, is a virtual assistant capable of understanding the questions of natural language doctors and providing an answer by specifying the source of information used. This device also allows you to photograph a prescription and analyze it automatically to detect potential drug interactions.
  The Synapse platform offers a panel of functions to help the doctor to prescribe medication.
  Arms: Assistance device

SUMMARY:
Polypharmacy in the older adults is common and promotes the risk of drug interactions. The hypothesis evoked is that a virtual platform with artificial intelligence applied to the health, and in particular to the good use of the drug, could bring aids to the doctors them of the prescription of drugs. The main objective of this study is to evaluate the impact of geriatric use of the Synapse platform on the frequency of inappropriate medication prescriptions (STOPP criteria) in discharge orders for patients 65 years of age or older hospitalized in geriatric department.

DETAILED DESCRIPTION:
The French 2018-2022 National Health Strategy plan aims to reduce the proportion of potentially harmful medication use. One particular challenge is the phenomenon of polypharmacy and inappropriate medication use in elderly, which is associated to an increased risk of drug-drug interactions. Several scales and tools have been proposed to identify inappropriate drugs prescription in older adults. Among them, the STOPP / START criteria (Screening Tool of Older Persons' Prescriptions / Screening Tool to Alert to Right Treatment) are internationally recognized.

The Synapse platform offers a panel of functions that may help physicians to prescribe medications. For instance, the prescriber can interact with the Synapse platform by asking any type of question about a drug (dosage, contraindication, interaction ...) before prescription. It also allows them to take a picture of prescription. The software detects in less than 10 seconds criteria for inappropriate medication prescriptions and potential drug-drug interactions.

More precisely, the Synapse platform provides information on a particular drug or prescription analysis regarding:

* Indications, contraindications, dosage and adverse effects of drugs.
* STOPP criteria.
* START criteria.
* Associations at risk for drug-drug interactions.

Multiple new health technologies are emerging, but few of them have demonstrated their scientific and medical added value using an evidence-based medicine approach.

This clinical trial aims to validate the clinical interest of the Synapse application in a geriatric environment.

Prescriptions made by geriatricians participating in this study will be analyzed by two independent experts, including one pharmacist and one geriatrician.

ELIGIBILITY:
* Inclusion criteria:

  * Male or female age aged more than 65 years
  * Hospitalization in geriatric department at Bordeaux University Hospital or Libourne Hospital
  * Initial drug prescription with at least 2 active pharmaceutical ingredients
  * Affiliation to French social security
  * Written informed consent signed by participant and investigator
* Exclusion criteria:

  * Adults protected by law
  * Subject included in a clinical trial with an experimental treatment
  * Subject during exclusion period relative to another trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with decrease in STOPP criteria number between initial prescription and exist prescription. | Month 6
  Proportion of patients with decrease in STOPP criteria number between initial prescription and exist prescription.

SECONDARY OUTCOMES:
Number of patients with increase in START criteria number between initial prescription and exist prescription. | Day 1
  Proportion of patients with increase in START criteria number between initial prescription and exist prescription.
Number of patients with increase in START criteria number between initial prescription and exist prescription. | Month 6
  Proportion of patients with increase in START criteria number between initial prescription and exist prescription.
Number of STOPP criteria | Day 1
  Difference in the number of STOPP criteria between initial and discharge prescription
Number of STOPP criteria | Month 6
  Difference in the number of STOPP criteria between initial and discharge prescription
Number of START criteria | Day 1
  Difference in the number of START criteria between initial and discharge prescription.
Number of START criteria | Month 6
  Difference in the number of START criteria between initial and discharge prescription.
number of patients with decrease in contraindicated drug-drug interaction | Day 1
  Proportion of patients with decrease in contraindicated drug-drug interaction number between initial and discharge prescription
number of patients with decrease in contraindicated drug-drug interaction | Month 6
  Proportion of patients with decrease in contraindicated drug-drug interaction number between initial and discharge prescription
Number of patients with decrease if active pharmaceutical ingredients | Day 1
  Proportion of patients with decrease in number of active pharmaceutical ingredients between initial and discharge prescription
Number of patients with decrease if active pharmaceutical ingredients | Month 6
  Proportion of patients with decrease in number of active pharmaceutical ingredients between initial and discharge prescription
Number of connections per week on Synapse platform by geriatricians | Month 6
  Number of connections per week on Synapse platform by geriatricians

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Olivier GIRODET, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (4):
- France (4):
  - CHU de Bordeaux, Hôpital Pellegrin, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier de Libourne - Pôle Gériatrie, Libourne
  - CHU de Bordeaux, Hôpital Xavier Arnozan, Pessac

IPD SHARING:
Plan to Share IPD: No